CLINICAL TRIAL: NCT04064346
Title: A Phase 3 Study of the Efficacy and Safety of Lixivaptan in Participants With Autosomal Dominant Polycystic Kidney Disease Consisting of a 1-year Double-blind, Placebo-controlled, Randomized Phase and a 1-year Open-label Phase: The ACTION Study
Brief Title: Efficacy and Safety of Lixivaptan in the Treatment of Autosomal Dominant Polycystic Kidney Disease
Acronym: ACTION
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The decision is based on a thorough reassessment of the commercial potential of lixivaptan as a potential best-in-class therapy for patients with autosomal dominant polycystic kidney disease (ADPKD).
Sponsor: Palladio Biosciences (Industry)
Collaborators: Centessa Pharmaceuticals plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA-ADPKD-301
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Results first posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Autosomal Dominant Polycystic Kidney; ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — lixivaptan

STUDY DESIGN:
Intervention Model Description: Part 1: 1-week, single-blind, Placebo Run-in Period, followed by a 5- to 6-week single-blind Lixivaptan Titration Period, followed by a 52-week Double-blind, Randomized Treatment Period, with 2/3 participants randomized to receive lixivaptan, and 1/3 participants randomized to receive placebo (the parallel assignment part of the study). There will be a 28-day off-treatment period during which final assessments will be obtained over 3 visits starting on the 8th day after the last dose of double-blind study drug through the 28th day after the last dose of double-blind study drug.
  Part 2: 2- to 4-week Lixivaptan Re-titration Period, followed by a 52-week Maintenance Treatment Period. There will be a 28-day off-treatment period during which final assessments will be obtained over 3 visits starting on the 8th day after the last dose of study drug through the 28th day after the last dose of study drug.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor - identical appearing active and placebo capsules in Part 1; all active capsules in Part 2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lixivaptan (Experimental): Lixivaptan capsules, 100-200 mg twice a day (BID)
  Interventions: Drug: Lixivaptan
- Placebo (Placebo Comparator): Matching placebo capsules BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lixivaptan — Oral vasopressin V2 receptor antagonist
  Arms: Lixivaptan
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 3 trial consisting of a 2-arm, double-blind, placebo-controlled, randomized phase (Part 1) followed by a single-arm open-label phase (Part 2) to demonstrate the efficacy and safety of lixivaptan in participants with autosomal dominant polycystic kidney disease (ADPKD). Part 1 of the trial is designed to demonstrate the efficacy of lixivaptan in slowing the decline in kidney function as measured by the difference in estimated glomerular filtration rate (eGFR) between the lixivaptan-treated and placebo-treated participants. Part 2 of the study is designed to provide confirmation of the durability of this effect. Additionally, both parts of the study will contribute to understanding the safety of lixivaptan, particularly any effects on liver chemistry tests.

DETAILED DESCRIPTION:
Part 1: Approximately 2250 participants with ADPKD will be screened in order to qualify the 1350 individuals who will proceed through the Placebo Run-in Period, the Lixivaptan Titration Period, and then be randomized to receive lixivaptan or placebo in the Double-blind, Randomized Treatment Period. Throughout Part 1 the study drug will look identical regardless of whether it is placebo or lixivaptan.

After meeting entry criteria during screening, participants will enter a 1-week single-blind, Placebo Run-in Period to obtain select baseline measurements. This will be followed by a 5- to 6-week single-blind dose titration period during which lixivaptan administered twice daily (BID) will be titrated to the highest tolerated dose (the Lixivaptan Titration Period). The starting dose (Level 1) will be 50 mg BID) and this will be increased weekly through Levels 2 (100 mg BID), 3 (150mg BID), and 4 (200 mg BID). The minimum dose to enter the next period, the Double-blind, Randomized Treatment Period, is Level 2 (100 mg BID). Those participants successfully titrated and tolerating the drug will then be randomized (each participant has a 2/3 chance of receiving lixivaptan and a 1/3 chance of receiving placebo) to either continue receiving lixivaptan or switch immediately to matching placebo in a double-blind manner. All dosing throughout the study will be 4 capsules BID. Depending on the study period, treatment arm to which the participant is randomized, and current dose level, the set of 4 capsules may be all placebo, all active or a combination of active and placebo. Double-blind treatment will continue for 52 weeks after which study drug will be held, and final assessments obtained off-treatment over 3 visits starting on the 8th day after the last dose of double-blind study drug through the 28th day after the last dose of study drug.

For Part 1 summaries after randomization, the analysis results will be presented by 2 treatment groups: lixivaptan and placebo.

Part 2: All participants entering Part 1, who have not discontinued due to an adverse event or withdrawn consent, will continue into Part 2 of the study, and will proceed through the Lixivaptan Re-titration Period and a Maintenance Treatment Period.

The Lixivaptan Re-titration Period will be a 2- to 4-week period during which dosing with lixivaptan will start at Level 1 (50 mg BID) for all participants and will be increased weekly until the dose level of lixivaptan, or the inferred lixivaptan dose level for participants randomized to placebo treatment, taken at the end of the Double-blind, Randomized Treatment Period in Part 1 is achieved. Lixivaptan treatment will continue for 52 weeks during the Maintenance Treatment Period after which study drug will be held, and final assessments obtained off-treatment over 3 visits starting on the 8th day after the last dose of lixivaptan through the 28th day after the last dose of lixivaptan.

Since all participants in Part 2 are treated with lixivaptan, the summaries for Part 2 will be presented in the following treatment cohorts and overall (treatment cohorts combined):

* Part1/Part2 - placebo/lixivaptan: all participants in Part 2 who were randomized into the placebo treatment group in Part 1.
* Part1/Part2 - lixivaptan/lixivaptan: all participants in Part 2 who were randomized into the lixivaptan treatment group in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADPKD by appropriate imaging or genetic testing.
* Mayo Clinic MRI imaging classification of 1C, 1D or 1E.
* eGFR ≥25 mL/min/1.73 m2 and ≤90 mL/min/1.73 m^2.
* Body mass index between 18 and 40 kg/m^2.
* Control of hypertension consistent with the 2021 Kidney Disease: Improving Global Outcomes guidelines without a diuretic and with an angiotensin converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB) unless not considered medically appropriate.
* Willing to practice acceptable methods of birth control (both males who have partners of child-bearing potential and females of childbearing potential).
* Able to provide informed consent.

Exclusion Criteria:

* Known sensitivity or idiosyncratic reaction to lixivaptan and/or its excipients.
* Hypovolemia.
* Abnormal serum sodium concentration at Screening.
* Subjects who have taken any investigational drug or used an investigational device within 30 days, or 5 half-lives, whichever is longer, prior to Screening.
* Subjects who are taking, have taken within the past 2 weeks, or are expected to be taking, strong or moderate CYP3A4 or CYP2C8 inhibitors or inducers including regular use of grapefruit juice or Seville oranges.
* Prior use of tolvaptan or lixivaptan within the past 2 months.
* Prior use of conivaptan, somatostatin analogs (e.g., lanreotide, pasireotide, octreotide, etc.), metformin, nicotinamide, bardoxolone, demeclocycline, or mammalian target of rapamycin kinase inhibitors (e.g., everolimus, sirolimus, etc.), or KetoCitra™ or any beta-hydroxybutyrate containing supplements to treat ADPKD within the past 2 months.
* Prior use of a sodium-glucose cotransporter 2 (SGLT2) inhibitor (e.g., canagliflozin, dapagliflozin, empagliflozin, etc.) within the past 2 months or expected need for initiation of treatment with a SGLT2 inhibitor during the study.
* Prior use of a hypoxia-inducible factor prolyl hydroxylase (HIF-PH) inhibitor within the past 2 months or expected need for initiation of treatment with a HIF-PH inhibitor during the study.
* Requirement for ongoing diuretic use.
* Advanced diabetes (e.g., glycosylated hemoglobin >7.5%, and/or glycosuria by dipstick, significant proteinuria [>300 mcg albumin/mg creatinine]), other significant kidney disease, kidney cancer, transplanted kidney, single kidney, recent kidney surgery within the past 6 months (including cyst drainage or fenestration) or acute kidney injury within past 6 months.
* Clinically significant incontinence, overactive bladder, or urinary retention (e.g., benign prostatic hyperplasia).
* New York Heart Association Functional Class 3 or 4 heart failure or other significant cardiac or ECG findings that could pose a safety risk to the subject.
* Positive test results for hepatitis B surface antigen or hepatitis C antibody.
* History of infection with human immunodeficiency virus unless the participant is clinically stable and doing well on a non-CYP interacting anti-retroviral therapy (ART) regimen and who has not required more than 2 changes in their ART regimen since treatment inception.
* History of clinically significant drug or alcohol abuse in the past 2 years.
* Contraindications to or interference with MRI assessments.
* Malignancy within the past 5 years except for those not considered to affect participant survival.
* Medical history or findings that preclude safe participation in the trial or participants who are likely to be non-compliant with trial procedures in the opinion of the Investigator or medical monitor.
* Clinically significant liver disease or impairment or alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin values >1.2 x ULN during Screening. Note: This criterion will preliminarily be reviewed at Visit 2 based on Visit 1a and Visit 1b results (if Visit 1b is required). The criterion must be re-evaluated no later than Visit 3 when results for Visit 2 are available.
* Simvastatin at a total daily dose >10 mg or amlodipine at a total daily dose >5 mg.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Torres, MD, PhD, Principal Investigator — Mayo Clinic
Locations (43):
- United States (23):
  - Nephrology Associates, PC - Greystone, Hoover, Alabama
  - Nephrology Consultants, LLC, Huntsville, Alabama
  - Arizona Kidney Disease & Hypertension Center - Scottsdale / Pima, Scottsdale, Arizona
  - JEM Research Institute, Atlantis, Florida
  - Elixia at Florida Kidney Physicians - Southeast, Fort Lauderdale, Florida
  - Qway Research, Hialeah, Florida
  - South Florida Nephrology Associates PA, Lauderdale Lakes, Florida
  - Total Research Group, LLC, Miami, Florida
  - Innovation Medical Research Center, Inc, Palmetto Bay, Florida
  - Florida Kidney Physicians - Tampa, Tampa, Florida
  - Clinical Site Partners, LLC, Winter Park, Florida
  - Tufts Medical Center, Inc,, Boston, Massachusetts
  - St Clair Nephrology Research, LLC, Roseville, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Angel City Research, Inc, Morrisville, North Carolina
  - Northeast Clinical Research Center, LLC, Bethlehem, Pennsylvania
  - Brown Medicine - Brown Physicians Patient Center, Riverside, Rhode Island
  - Knoxville Kidney Center LLC, Knoxville, Tennessee
  - Prolato Clinical Research Center (PCRC), Houston, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - Utah Kidney Research Institute, Salt Lake City, Utah
  - Nephrology Associates of Northern Virginia, Inc, Fairfax, Virginia
- Renal Research - Gosford, Gosford, New South Wales, Australia
- Bulgaria (5):
  - University Multiprofile Hospital for Active Treatment, Pleven
  - University Multiprofile Hospital for Active Treatment - Kaspela, Plovdiv
  - Medical Center "Hipokrat - N", Plovdiv
  - Kidney Center - Medical Center, Varna
  - Multi-Profile Hospital for Active Treatment Sveta Anna - Varna, Varna
- Hungary (5):
  - Bajai Szent Rokus Korhaz, Baja
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem, Debrecen
  - Bugat Pal Korhaz, Gyöngyös
  - University of Pecs, Pécs
- Poland (2):
  - SCM Spolka z o.o, Krakow
  - Provita Centrum Medyczne sp. z o.o., Warsaw
- Spain (2):
  - Hospital Universitari de Bellvitge (HUB), Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
- Turkey (Türkiye) (4):
  - T.R. Ministry of Health Ankara Training and Research Hospital (Internal Disease, Division of Nephrology), Ankara
  - Bezmialem Vakif Universitesi Tip Fakultesi Hastanesi, Fatih
  - Istanbul Universitesi - Cerrahpasa Tip Fakultesi Hastanesi (IUCTFH), Fatih
  - Erciyes Universitesi Tip Fakultesi (Erciyes University Faculty of Medicine) (Internal Medicine; Nephrology), Kayseri
- Salford Royal NHS Foundation Trust, Salford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects Pre-randomization: After meeting entry criteria during screening, the single-blind pre-randomization period (up to 7 weeks) consisted of:
  1. A 1-week single-blind, Placebo Run-in Period during which participants self-administered 4 capsules containing placebo twice daily for 1 week.
  2. A 5- to 6-week single-blind dose titration period during which lixivaptan administered twice daily (BID) was titrated to the highest tolerated dose (the Lixivaptan Titration Period).
- Lixivaptan: Randomized Double-blind Period (52 weeks):
  Participants in this group successfully titrated and tolerated the drug were randomized to continue receiving lixivaptan at the dose level achieved at the end of the Lixivaptan Titration Period.
- Placebo: Randomized Double-blind Period (52 weeks):
  Participants in this group successfully titrated and tolerated the drug were randomized to receive placebo matched to the dose level of lixivaptan achieved at the end of the Lixivaptan Titration Period.
Period: Pre-randomization Single-blind Period
Arm/Group | All Subjects Pre-randomization | Lixivaptan | Placebo
Started | 12 | 0 (This arm was not applicable for the Pre-randomization Single-blind Period.) | 0 (This arm was not applicable for the Pre-randomization Single-blind Period.)
Treated in Placebo Run-in | 12 | 0 | 0
Treated in Lixivaptan Titration Period | 8 | 0 | 0
Completed | 5 | 0 | 0
Not Completed | 7 | 0 | 0
Period: Randomized Double-blind Period
Arm/Group | All Subjects Pre-randomization | Lixivaptan | Placebo
Started | 0 (This arm was not applicable for the Randomized Double-blind Period.) | 4 | 1
Randomized | 0 | 4 | 1
Completed | 0 | 4 (1 participant withdrew consent before entering Follow-up Period I.) | 1
Not Completed | 0 | 0 | 0
Period: Follow-up Period I
Arm/Group | All Subjects Pre-randomization | Lixivaptan | Placebo
Started | 0 (This arm was not applicable for Follow-up Period I.) | 3 (1 participant who completed the Randomized Double-blind Period withdrew consent before entering Follow-up Period I.) | 1
Completed | 0 | 3 (The study was terminated prematurely before any participants proceeded to the Re-titration Period.) | 1 (The study was terminated prematurely before any participants proceeded to the Re-titration Period.)
Not Completed | 0 | 0 | 0
Period: Re-titration Period
Arm/Group | All Subjects Pre-randomization | Lixivaptan | Placebo
Started | 0 (This arm was not applicable for the Re-titration Period.) | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Maintenance Treatment Period
Arm/Group | All Subjects Pre-randomization | Lixivaptan | Placebo
Started | 0 (This arm was not applicable for the Maintenance Treatment Period.) | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Follow-up Period II
Arm/Group | All Subjects Pre-randomization | Lixivaptan | Placebo
Started | 0 (This arm was not applicable for Follow-up Period II.) | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Participants: The baseline population consisted of all enrolled participants.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.9 (8.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
  Bulgaria | 2
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.47 (6.795)
Family History of Autosomal Dominant Polycystic Kidney Disease [Count of Participants; unit: Participants]
  Yes | 10
  No | 2

OUTCOME MEASURES:

1. Primary Outcome: Annualized Change in Estimated Glomerular Filtration Rate (eGFR) - Part 1
Description: The annualized change in eGFR will be calculated from the Chronic Kidney Disease Epidemiology Collaboration eGFR creatinine equation refit without the race variable (CKD-EPIcr_R) equation for serum creatinine from baseline (mean of 3 eGFR determinations obtained during Screening and Placebo Run-in Periods [Visits 1a/1b (if required), Visit 2, and Visit 3]) to final assessment (mean of 3 eGFR determinations obtained during Follow-up Period I or, for participants who discontinue treatment prior to Visit 22, during the Follow-up Period 8 to 28 days following study drug treatment discontinuation).
Time Frame: Baseline to the end of Follow-up Period I (up to 71 weeks)
Population: Efficacy data were not analyzed as only 5 participants were randomized, and all 5 participants were prematurely terminated from the study drug by the sponsor less than 1 month following randomization. One month after randomization was the first scheduled post-randomization visit during which efficacy parameters would have been collected.
Arm/Group | Lixivaptan | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Annualized Change in Estimated Glomerular Filtration Rate (eGFR) - Part 2
Description: The annualized change in eGFR will be calculated from the CKD-EPIcr_R equation for serum creatinine from baseline (mean of 3 eGFR determinations obtained during obtained during Follow-up Period I) to final assessment (mean of 3 eGFR determinations obtained during Follow-up Period II or, for participants who discontinue treatment prior to Visit 43, during the Follow-up Period 8 to 28 days following study drug treatment discontinuation).
Time Frame: Baseline to the end of Follow-up Period II (up to 64 weeks)
Population: Efficacy data were not analyzed as only 5 participants were randomized, and all 5 participants were prematurely terminated from the study drug by the sponsor less than 1 month following randomization. One month after randomization was the first scheduled post-randomization visit during which efficacy parameters would have been collected. The study terminated prior to any participants entering Part 2 of study.
Groups:
- Randomized to Lixivaptan in Part 1: All participants who were randomized to treatment with lixivaptan in the Randomized Double-blind Period in Part 1 and were to receive lixivaptan in Part 2.
- Randomized to Placebo in Part 1: All participants who were randomized to treatment with placebo in the Randomized Double-blind Period in Part 1 and were to receive lixivaptan in Part 2.
Arm/Group | Randomized to Lixivaptan in Part 1 | Randomized to Placebo in Part 1
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Serum Alanine Aminotransferase (ALT) Levels >3 × the Upper Limit of Normal (ULN) - Part 1
Description: Number of participants randomized to lixivaptan with serum ALT levels >3 × the ULN compared to those randomized to placebo. The normal range of ALT was defined as 0-33 or 0-44 U/L, depending on the lab used.
Time Frame: From the end of the Single-blind Lixivaptan Titration Period to the end of Follow-up Period I (maximum of 102 days)
Population: All participants who entered the Double-blind Randomized Treatment Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Lixivaptan | Placebo
Number analyzed (Participants) | 4 | 1
Participants | 0 | 1

4. Secondary Outcome: Number of Participants With Serum ALT Levels >3 × the ULN - Part 2
Description: Number of participants randomized to lixivaptan with serum ALT levels >3 × ULN compared to those randomized to placebo. The normal range of ALT was defined as 0-33 or 0-44 U/L, depending on the lab used.
Time Frame: Duration of the Lixivaptan Re-titration Period and the Maintenance Treatment Period (56 weeks) and Follow-up Period II (4 weeks)
Population: The study terminated prior to any participants entering Part 2 of study.
Arm/Group | Randomized to Lixivaptan in Part 1 | Randomized to Placebo in Part 1
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: eGFR Slope - Part 1
Description: Annualized rate of change (slope) in eGFR for serum creatinine, based on all eGFR determinations from baseline to all visits with on-treatment eGFR values during the Double-blind, Randomized Treatment Period. The baseline value will be calculated as the mean of 3 eGFR determinations obtained during Screening and Placebo Run-in Periods (Visits 1a/1b [if required], Visit 2, and Visit 3).
Time Frame: Baseline to the end of Double-blind Randomized Treatment Period (up to 67 weeks), with changes from baseline calculated every 4 weeks during the Double-blind Randomized Treatment Period
Population: as for outcome 1
Arm/Group | Lixivaptan | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: eGFR Slope - Part 2
Description: Annualized rate of change (slope) in eGFR for serum creatinine, based on all eGFR determinations from baseline to all visits with on-treatment eGFR values during the Maintenance Treatment Period. The baseline value will be calculated as the mean of 3 eGFR determinations obtained during obtained during Follow-up Period I.
Time Frame: Baseline to the end of the Maintenance Treatment Period (up to 60 weeks), with changes from baseline calculated every 4 weeks during the Maintenance Treatment Period
Population: as for outcome 2
Arm/Group | Randomized to Lixivaptan in Part 1 | Randomized to Placebo in Part 1
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Height-adjusted Total Kidney Volume (htTKV) - Part 1
Description: Annualized percent change in htTKV, determined by magnetic resonance imaging (MRI), from baseline (obtained at Screening [Visit 1a]) to the end of Follow-up Period I.
Time Frame: Baseline to the end of Follow-up Period I (up to 71 weeks)
Population: as for outcome 1
Arm/Group | Lixivaptan | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Height-adjusted Total Kidney Volume (htTKV) - Part 2
Description: Annualized percent change in htTKV, determined by MRI from baseline (obtained at Visit 25/Week 56) to the end of Follow-up Period II.
Time Frame: Baseline to the end of Follow-up Period II (up to 60 weeks)
Population: as for outcome 2
Arm/Group | Randomized to Lixivaptan in Part 1 | Randomized to Placebo in Part 1
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) During the Lixivaptan Titration Period in Part 1
Description: Number of participants with TEAEs during the Lixivaptan Titration Period.
Time Frame: Up to 6 weeks
Population: All participants entering the Lixivaptan Titration Period.
Measure: Count of Participants; unit: Participants
Groups:
- Lixivaptan Titration Period Participants: All participants who took at least one dose of lixivaptan during the Lixivaptan Titration Period in Part 1
Arm/Group | Lixivaptan Titration Period Participants
Number analyzed (Participants) | 8
Participants | 3

10. Secondary Outcome: Number of Participants With TEAEs After Randomization in Part 1
Description: Number of participants with TEAEs by treatment group after Randomization (Double-blind Randomized Treatment Period and Follow-up Period I)
Time Frame: From Randomization to study completion (up to 102 days)
Population: All participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Lixivaptan | Placebo
Number analyzed (Participants) | 4 | 1
Participants | 1 | 1

11. Secondary Outcome: Number of Participants With TEAEs in Part 2
Description: Number of participants with TEAEs by treatment cohort during Part 2 (Lixivaptan Re-titration Period, Maintenance Treatment Period, and Follow-up Period II).
Time Frame: Up to 60 weeks
Population: All participants were prematurely terminated from the study drug by the sponsor less than 1 month following randomization; none proceeded to Part 2 of the study.
Arm/Group | Randomized to Lixivaptan in Part 1 | Randomized to Placebo in Part 1
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants With Potentially Clinically Important Clinical Laboratory Findings During the Lixivaptan Titration Period in Part 1
Description: Number of participants with clinical laboratory findings (clinical chemistry, hematology and urinalysis) recorded during the Lixivaptan Titration Period and considered to be potentially clinically important.
Time Frame: Up to 6 weeks
Population: All participants entering the Lixivaptan Titration Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Lixivaptan Titration Period Participants
Number analyzed (Participants) | 8
Participants | 0

13. Secondary Outcome: Number of Participants With Potentially Clinically Important Clinical Laboratory Findings After Randomization in Part 1
Description: Number of participants with clinical laboratory findings (clinical chemistry, hematology and urinalysis) recorded after Randomization (Double-blind Randomized Treatment Period and Follow-up Period I) and considered to be potentially clinically important, by treatment group.
Time Frame: From Randomization to last clinical laboratory evaluation (up to 102 days)
Population: All participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Lixivaptan | Placebo
Number analyzed (Participants) | 4 | 1
Participants | 0 | 0

14. Secondary Outcome: Number of Participants With Potentially Clinically Important Clinical Laboratory Findings in Part 2
Description: Number of participants with clinical laboratory findings (clinical chemistry, hematology and urinalysis) recorded during Part 2 (Lixivaptan Re-titration Period, Maintenance Treatment Period, and Follow-up Period II) and considered to be potentially clinically important, by treatment cohort.
Time Frame: Up to 60 weeks
Population: as for outcome 11
Arm/Group | Randomized to Lixivaptan in Part 1 | Randomized to Placebo in Part 1
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Number of Participants With Potentially Clinically Important Vital Signs Findings During the Lixivaptan Titration Period in Part 1
Description: Number of participants with vital signs findings (heart rate, diastolic and systolic blood pressure, weight) recorded during the Lixivaptan Titration Period and considered to be potentially clinically important.
Time Frame: Up to 6 weeks
Population: All participants entering the Lixivaptan Titration Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Lixivaptan Titration Period Participants
Number analyzed (Participants) | 8
Participants | 0

16. Secondary Outcome: Number of Participants With Potentially Clinically Important Vital Signs Findings After Randomization in Part 1
Description: Number of participants with vital signs findings (heart rate, diastolic and systolic blood pressure, weight) recorded after Randomization (Double-blind Randomized Treatment Period and Follow-up Period I) and considered to be potentially clinically important, by treatment group.
Time Frame: From Randomization to last measurement of vital signs (up to 102 days)
Population: All participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Lixivaptan | Placebo
Number analyzed (Participants) | 4 | 1
Participants | 0 | 0

17. Secondary Outcome: Number of Participants With Potentially Clinically Important Vital Signs Findings in Part 2
Description: Number of participants with vital signs findings (heart rate, diastolic and systolic blood pressure, weight) recorded during Part 2 (Lixivaptan Re-titration Period, Maintenance Treatment Period, and Follow-up Period II) and considered to be potentially clinically important, by treatment cohort.
Time Frame: Up to 60 weeks
Population: as for outcome 11
Arm/Group | Randomized to Lixivaptan in Part 1 | Randomized to Placebo in Part 1
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Number of Participants With Potentially Clinically Significant 12-lead Electrocardiogram (ECG) Findings During the Lixivaptan Titration Period in Part 1
Description: Number of participants with ECG findings recorded during the Lixivaptan Titration Period and considered to be potentially clinically important (defined as a QT interval corrected for heart rate according to Fridericia's formula [QTcF] ≥ 450 msec).
Time Frame: Up to 6 weeks
Population: All participants entering the Lixivaptan Titration Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Lixivaptan Titration Period Participants
Number analyzed (Participants) | 8
Participants | 0

19. Secondary Outcome: Number of Participants With Potentially Clinically Significant 12-lead ECG Findings After Randomization in Part 1
Description: Number of participants with ECG findings recorded after Randomization (Double-blind Randomized Treatment Period and Follow-up Period I) and considered to be potentially clinically important (defined as a QTcF ≥ 450 msec), by treatment group.
Time Frame: From Randomization to last ECG (up to 102 days)
Population: All participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Lixivaptan | Placebo
Number analyzed (Participants) | 4 | 1
Participants | 0 | 0

20. Secondary Outcome: Number of Participants With Potentially Clinically Significant 12-lead ECG Findings in Part 2
Description: Number of participants with ECG findings recorded during Part 2 (Lixivaptan Re-titration Period, Maintenance Treatment Period, and Follow-up Period II) and considered to be potentially clinically important (defined as a QTcF ≥ 450 msec), by treatment cohort.
Time Frame: Up to 60 weeks
Population: as for outcome 11
Arm/Group | Randomized to Lixivaptan in Part 1 | Randomized to Placebo in Part 1
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from when participants had taken their first dose of lixivaptan in the Lixivaptan Titration Period until the end of the study (maximum duration: 123 days)
Groups:
- Lixivaptan Titration Period: All participants who took at least one dose of lixivaptan during the Lixivaptan Titration Period in Part 1
- Lixivaptan (Randomized Treatment Period): Lixivaptan capsules, 100-200 mg twice a day (BID)
  Lixivaptan: Oral vasopressin V2 receptor antagonist
- Placebo (Randomized Treatment Period): Matching placebo capsules BID
  Placebo: Matching placebo
Arm/Group | Lixivaptan Titration Period | Lixivaptan (Randomized Treatment Period) | Placebo (Randomized Treatment Period)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 3/8 | 1/4 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lixivaptan Titration Period (N=8) | Lixivaptan (Randomized Treatment Period) (N=4) | Placebo (Randomized Treatment Period) (N=1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal cyst ruptured (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT04064346/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT04064346/SAP_001.pdf